CLINICAL TRIAL: NCT04385524
Title: Use of Dynavax Heplisav B in Healthcare Workers Previously Vaccinated With Standard 3-dose Vaccine Who Failed to Demonstrate Seroprotection
Brief Title: Use of Dynavax Heplisav B in Healthcare Workers Previously Vaccinated With 3-dose Vaccine Who Failed to Demonstrate Seroprotection
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: We decided to close this study. We are unable to perform this study due to the current pandemic.
Sponsor: University of Louisville (Other)
Collaborators: Dynavax Technologies Corporation (Industry)
Responsible Party: Principal Investigator, Ruth Carrico, Professor, University of Louisville
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 191219
Record Dates: First submitted 2019-12-10; First posted 2020-05-13 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Hepatitis B Virus
Keywords: Hepatitis B vaccine; Hepatitis B vaccine non-responder; Hepatitis B seroconversion
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Vaccination (Other): Heplisav B vaccine will be administered to subjects demonstrating completion of two prior series of standard 3-dose Hepatitis B vaccine but still without evidence of seroconversion.
  One dose (20 mcg) of vaccine will be administered intramuscularly followed by Hepatitis B quantitative antibody titer 30-60 days later.
  If still Hepatitis B antibody negative, a second dose (20 mcg) of vaccine will be administered intramuscularly followed by a Hepatitis B quantitative titer 30-60 days later.
  If still no evidence of Hepatitis B immunity (10iU antibody or greater), will be deemed a non-responder to this vaccine
  Interventions: Biological: Adjuvanted Hepatitis B Vaccine

INTERVENTIONS:
Biological: Adjuvanted Hepatitis B Vaccine — Adjuvanted Hepatitis B vaccine will be provided to healthcare workers previously vaccinated with the standard 3-dose series of Hepatitis B vaccine but who have failed to respond to two complete 3-dose series

SUMMARY:
Protection against Hepatitis B infection is a regulatory and safety cornerstone to infection prevention and control programs involving the healthcare workforce in the United States. Until 2018 when a new adjuvanted vaccine was released, immunization for this population has involved a three-dose series followed by an additional three-dose series for those demonstrating lack of seroprotection. If that lack continued following the second three-dose series, and verification of a negative Hepatitis B antigen status, that person has historically been deemed a non-responder to Hepatitis B vaccine and at potential risk for infection. This non-response status may be used to determine job responsibilities representing excessive risk for the healthcare worker resulting in potential career and practice limitations and decisions. With the release of the new adjuvanted vaccine, there is potential to determine the role that new vaccine may play in promoting an immune response among this non-responding subset of at-risk healthcare workers. The aims of this study include: 1) determining the effect of this adjuvanted vaccine in producing seropositivity in a population of healthcare personnel previously deemed as non-responders following administration of two rounds of the traditional 3-dose series of Hepatitis B vaccine and confirmation of negative Hepatitis B antigen; and 2) determining the personal and professional impact of the lack of immunity to Hepatitis B among healthcare personnel.

DETAILED DESCRIPTION:
Background Protection against Hepatitis B infection is a regulatory and safety cornerstone to infection prevention and control programs involving the healthcare workforce in the United States. Until 2018 when a new adjuvanted vaccine was released, immunization for this population has involved a three-dose series followed by an additional three-dose series for those demonstrating lack of seroprotection. If that lack continued following the second three-dose series, and verification of a negative Hepatitis B antigen status, that person has historically been deemed a non-responder to Hepatitis B vaccine and at potential risk for infection. This non-response status may be used to determine job responsibilities representing excessive risk for the healthcare worker resulting in potential career and practice limitations and decisions. With the release of the new adjuvanted vaccine, there is potential to determine the role that new vaccine may play in promoting an immune response among this non-responding subset of at-risk healthcare workers.

Heplisav B is a standard of care vaccine that provides an alternative to a traditional 3-dose series by enabling use of a 2-dose series with doses one and two separated by one month. Work by Jackson and Janssen have indicated a greater than 90% seroprotection, perhaps closer to 100%, with the 2-dose series of this adjuvanted vaccine where hyporesponsiveness to 3-dose vaccines has been noted, principally in persons who smoke, are diabetic, obese, and male. This shorter administration schedule and reduced number of doses, combined with the seroconversion data make this vaccine ideal for situations where rapid induction of immunization occurs, such as those working in exposure-risk jobs such as healthcare.

The aims of this study include: 1) determining the effect of this adjuvanted vaccine in producing seropositivity in a population of healthcare personnel previously deemed as non-responders following administration of two rounds of the traditional 3-dose series of Hepatitis B vaccine and confirmation of negative Hepatitis B antigen; and 2) determining the personal and professional impact of the lack of immunity to Hepatitis B among healthcare personnel.

Use of Heplisav B will follow the FDA labeling and will not involve off-label use. Study personnel will work with the employee/occupational health and infection control departments to identify healthcare personnel working in a Louisville hospital, long term care facility, or clinic meeting the definition of a non-responder. Work will be done with University of Louisville Campus Health Services leadership to identify students, residents, fellows, or faculty who meet the definition of a non-responder. After gaining consent for participation in the study, titers will be drawn to document current Hepatitis B quantitative antibody and antigen levels. Enrolled participants (those with negative antibody and antigen) will be administered one dose of the adjuvanted vaccine followed by repeat antigen and antibody testing 30-60 days after receipt of that dose of vaccine. If results of the antibody and antigen are again negative, a second dose of the adjuvanted vaccine will be administered followed by repeat antibody and antigen testing 30-60 days after receipt of that dose of vaccine. For those healthcare personnel enrolled in the study, a questionnaire will be administered designed to understand the personal and professional impact of a non-responder status to hepatitis B.

All doses of Heplisav B vaccine will be provided by Dynavax and will be at no cost to the participants. All labs drawn will also be at no cost to the participant.

Study participants will be seen for a total of up to 9 visits with participation in the study lasting approximately 3 months. Visits involving labwork, vaccine administration, and the survey will occur in-person at the University of Louisville International Travel Clinic located in MedCenter One (501 East Broadway, Louisville Kentucky 40202). Visits gathering information regarding adverse reactions to vaccination will occur via telephone call visits as well as during in-person visits after the vaccine dose(s) have been administered.

ELIGIBILITY:
Inclusion Criteria:

Healthcare personnel age 18-64 years of age who have documentation of prior receipt of two rounds of the traditional 3-dose series of Hepatitis B vaccine and having serologic testing demonstrating quantitative Hepatitis B antibody level of less than 10 iU and a negative Hepatitis B antigen.

Exclusion Criteria:

1. Pregnancy
2. Allergy to the adjuvanted vaccine or a vaccine component
3. Sensitivity to yeast
4. Persons unable to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2021-02-01 (Estimated); Study Completion 2021-02-28 (Estimated)

PRIMARY OUTCOMES:
Hepatitis B Seroconversion as Measured by Achievement of 10iU/ml on Quantitative Hepatitis B Titer | within 3 months of acceptance into the study
  Demonstration of Hepatitis B immunity via achievement of 10iU/ml or greater on quantitative titer following 1 or 2 doses of the adjuvanted Hepatitis B vaccine

SECONDARY OUTCOMES:
Reported Impact of Non-Response Status on Career and Personal Economics as Reported by Healthcare Worker | within 6 months of acceptance into the study
  Impact of Hepatitis B non-response status on career and personal economics as perceived by the healthcare worker completing the survey. This includes metrics such as hourly wage, job promotion, career pathway

IPD SHARING:
Plan to Share IPD: No